CLINICAL TRIAL: NCT01547507
Title: Performance Evaluation of AirWay Medix Closed Suction System Compared With a Standard Closed Suction System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biovo Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Biovo-12-CTIL
Record Dates: First submitted 2012-02-22; First posted 2012-03-08 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Endotracheal Tube; Mechanical Ventilation
Keywords: hemodynamics; respiratory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KimVent Turbo-Cleaning Closed Suction System Kimberly clark (Active Comparator)
  Interventions: Device: AirWay Medix Closed Suction System
- Airway Medix Closed Suction System (Active Comparator)
  Interventions: Device: AirWay Medix Closed Suction System

INTERVENTIONS:
Device: AirWay Medix Closed Suction System — AirWay Medix Closed Suction System

SUMMARY:
The aim of this prospective, randomized study is to compare the performance, safety, and ease of use (usability) between two closed suction systems, the AirWay Medix Closed Suction System and Kimberly KimVent while intubated with an endotracheal in hospitals and ICU. 26 adults with an endotracheal tube and mechanical ventilation will be randomized into 2 groups to receive one of the following closed suction systems endotracheal tubes:

1. AirWay Medix Closed Suction System
2. KimVent Turbo-Cleaning Closed Suction System Kimberly clarK The groups will be compared regarding the safety, performance and ease of use (usability).

ELIGIBILITY:
Inclusion Criteria:

1. Aged greater than 18 years
2. Mechanically ventilated for more than 6 hours
3. Endotracheal intubation anticipated to be routine (not difficult) based upon preoperative airway assessment
4. Signed informed consent
5. Sexually active female subjects of childbearing potential must be practicing adequate contraception during the treatment period -

Exclusion Criteria:

1. Gross / massive hemoptysis
2. Received lung transplantation in the past
3. Admitted from other hospital already mechanically ventilated
4. Previously received mechanical ventilation
5. Active bronchial bleeding
6. Pregnant women, women who plan to become pregnant and breastfeeding women.
7. Substance or alcohol abuse
8. Participation in concurrent trials
9. Any reasons making the patient a poor candidate in the opinion of the investigator -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
hemodynamic and respiratory data | Patients will be followed until extubation

CONTACTS AND LOCATIONS:
Overall Officials: Nimrod Adi, MD, Principal Investigator — Kaplan Medical Center
Locations (1):
- Kaplaan MC, Rehovot, Israel